CLINICAL TRIAL: NCT07128329
Title: The Acute Effects of Oral Nicotine Pouches Among Infrequent and Frequent Nicotine/Tobacco Users
Brief Title: Acute Effects of Oral Nicotine Pouches
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00502492; 5R01DA055962-04 (NIH)
Record Dates: First submitted 2025-08-13; First posted 2025-08-18 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Nicotine Pouch Self-Administration; Nicotine Pharmacokinetic Study; Nicotine Pharmacodynamic Study
Keywords: Nicotine pouch; Cigarette smokers; Infrequent nicotine users; Outpatient; Zyn

STUDY DESIGN:
Intervention Model Description: Mixed between/within-subjects crossover design with two groups of participants (cigarette smokers and infrequent nicotine users). Participants complete all experimental sessions, serving as their own control.
Who Masked: Participant, Outcomes Assessor
Masking Description: Research program coordinators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pouch label version 1 (Active Comparator): Nicotine pouches with label 1
  Interventions: Drug: Nicotine Pouches
- Pouch label version 2 (Experimental): Nicotine pouches with label 2
  Interventions: Drug: Nicotine Pouches

INTERVENTIONS:
Drug: Nicotine Pouches — Nicotine pouches
  Other Names: Zyn

SUMMARY:
The present human laboratory study will recruit cigarette smokers (n=60) and adult infrequent nicotine users (n=60) to complete two counterbalanced lab sessions in which the participants use nicotine pouches under controlled conditions. The investigators are recruiting both frequent and infrequent nicotine users because FDA regulates tobacco products based on a public health standard, meaning FDA must consider the impact a regulation may have on the population as a whole (e.g., people who use and do not use tobacco products currently).

DETAILED DESCRIPTION:
This study will be conducted at the Johns Hopkins Behavioral Pharmacology Research unit (BPRU). Participants will complete a screening visit, and, if eligible, will then complete 2 outpatient experimental sessions (separated by at least 48 hours). The study will use a mixed between/within-subjects crossover design. The between-subjects component is because there are two groups of participants (60 cigarette smokers, 60 infrequent nicotine users) and the within-subjects component is because participants complete all experimental sessions (thus, serving as the participant's own control). Smokers will be instructed to abstain from all tobacco 12 hours prior to each session so that the participants begin study sessions in a state of nicotine/tobacco withdrawal. Sessions will be completed in a counterbalanced order to reduce order effects. During each experimental session, a battery of assessments including subjective questionnaires (abuse liability, nicotine-related effects, withdrawal suppression), cognitive performance, blood collection for pharmacokinetic analysis (this will be optional), vital signs, and pouch use (or topography) will be conducted

ELIGIBILITY:
Inclusion criteria (all participants):

* greater than or equal to 21 years old
* good general health based on screening procedures
* vital signs in normal range (resting heart rate less than 110bpm, systolic blood pressure less than 150mmHg, diastolic blood pressure less than 100mmHg)
* negative urine test for illicit drug use (excluding THC) and negative breath alcohol test at screening and before each session
* no self-reported prior use of oral nicotine pouches
* Not actively trying to quit smoking or using smoking cessation medication (e.g., nicotine replacement therapy)

Additional inclusion criteria (smokers):

* self-report currently smoking cigarettes daily
* exhaled breath CO greater than or equal to 10ppm and urine cotinine greater than 100 ng/ml at screening
* meet criteria for tobacco use disorder
* no self-reported regular use of other tobacco products (e.g., smokeless products, e-cigarettes) in the past 30 days

Additional inclusion criteria (non-nicotine users):

* self-report previously using nicotine/tobacco but no more than 100 lifetime uses across all routes of administration
* no self-reported nicotine/tobacco uses in the past 30 days
* urine cotinine less than 100 ng/ml at screening.

Exclusion criteria (all participants):

* psychoactive drug use (aside from cannabis, nicotine, alcohol, or caffeine) in past month
* current use of OTC drugs, supplements/vitamins, or prescription medications that, in the opinion of medical staff, will impact safety
* currently have severe dependence for cannabis
* history of or current significant medical condition that, in the opinion of medical staff, will impact safety
* current psychiatric condition or substance use disorder (aside from tobacco use disorder for smokers), that, in the opinion of medical staff, will impact safety
* women who are pregnant, planning to become pregnant, or are breast-feeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics - CMax for nicotine | 6.5 hours
  Blood plasma samples will be collected and sent to a designated laboratory for quantitative analysis of nicotine. Maximum concentration (Cmax), is the highest plasma nicotine concentration reached during a session and provides important insight into the abuse liability of a tobacco product.
Pharmacokinetics - AUC for nicotine | 6.5 hours
  Blood plasma samples will be collected and sent to a designated laboratory for quantitative analysis of nicotine. Area under the curve (AUC), represents the total nicotine exposure during an entire session and provides important insight into the abuse liability of a tobacco product.
Drug Effect Questionnaire-Like Drug Effect | 6.5 hours
  The DEQ will be used to obtain subjective ratings of "like drug effect". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effect Questionnaire-pleasant Drug Effect | 6.5 hours
  The DEQ will be used to obtain subjective ratings of "pleasant drug effect". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effect Questionnaire-take again | 6.5 hours
  The DEQ will be used to obtain subjective ratings of "take again". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Topography - number of pouches used | 2 hours
  During the 2 hour ad libitum bout, primary topography variable will be collected - the total number of pouches used (range 0 - 5)
Topography - duration of use | 2 hours
  During the 2 hour ad libitum bout, primary topography variable will be collected - total duration of use (range 0 - 2 hours).
Hughes-Hatsukami Withdrawal Questionnaire | 6.5 hours
  The HHWS will be used to obtain subjective ratings of tobacco withdrawal outcomes among smokers including: "urge", "craving" "Anxious," "Depression," " Difficultly concentrating," "Drowsy," "Hunger," "Impatient," "Irritable," "Restlessness," "Desire for sweets". Scores for these items range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Tiffany-Drobes Questionnaire on Smoking Urges (QSU) brief | 6.5 hours
  The QSU-brief will measure tobacco withdrawal symptoms in smokers using 10 items that form 2 factors: factor 1 (intention to smoke) and factor 2 (anticipation of withdrawal symptom relief). Mean score 0-5. Lower score is better.

SECONDARY OUTCOMES:
Pharmacokinetics - Tmax for nicotine | 6.5 hours
  Blood plasma samples will be collected and sent to a designated laboratory for quantitative analysis of nicotine. Time to max concentration (Tmax), is the time (in min) to reach Cmax. This is another measure relevant for abuse liability. Range is 0 - 20 min for directed period
The Direct Effects of Nicotine Scale (DENS) | 6.5 hours
  The DENS will assess nicotine-specific effects via 10 items "Confused," "Dizzy," "Headache," "Heart Pound," "Lightheaded," "Nauseous," "Nervous," "Salivation," "Sweaty," and "Weak". Each item is scored separately from 0 (not at all) to 100 (extremely).
Drug Effects Questionnaire (DEQ) - feel drug effect | 6.5 hours
  The DEQ will assess subjective ratings for "feel drug effect". Scores range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effects Questionnaire (DEQ) subjective effects- unpleasant effect | 6.5 hours
  The DEQ will assess subjective ratings for "unpleasant drug effect". Scores range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effects Questionnaire (DEQ) subjective effects- dislike drug effect | 6.5 hours
  The DEQ will assess subjective ratings for "dislike drug effect". Scores range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.

CONTACTS AND LOCATIONS:
Overall Officials: Tory Spindle, PhD, Principal Investigator — Johns Hopkins University School of Medicine, Department of Psychiatry and Behavioral Sciences
Locations (1):
- Johns Hopkins University School of Medicine, Behavioral Pharmacology Research Unit (Bayview), Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No